CLINICAL TRIAL: NCT01910298
Title: A Prospective, Multicenter, Controlled Study of Implant-based Breast Reconstruction, Measuring the Safety, Efficacy and Outcomes, of Immediate Single Stage Breast Reconstruction With Strattice™ Reconstructive Tissue Matrix Versus Immediate Two Stage Breast Reconstruction Without Strattice™ TM (ESSBR-Efficacy of Single Stage Breast Reconstruction)
Brief Title: Efficacy Study of Single Stage Breast Reconstruction in Female Participants With Mastectomy
Acronym: ESSBR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is being terminated due to no enrollment in over one year in the control arm
Sponsor: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LFC 2012.06.01
Record Dates: First submitted 2013-07-22; First posted 2013-07-29 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-04

CONDITIONS: Mastectomy and Breast Reconstruction
Keywords: Breast reconstruction; Breast implant; Breast cancer; Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty; Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breast Reconstruction, Direct to Implant (DTI) with Strattice™ (Active Comparator): Participants underwent immediate post-mastectomy breast reconstruction with a breast implant and Strattice™ reconstructive tissue matrix (surgical mesh).
  Interventions: Procedure: Breast Reconstruction, Direct to Implant (DTI) with Strattice™
- Two Stage Breast Reconstruction (Active Comparator): Participants underwent immediate, two-stage post-mastectomy breast reconstruction without reinforcement. Initial placement of a tissue expander that was inflated for approximately one to six months, and then replaced with an implant.
  Interventions: Procedure: Two Stage Breast Reconstruction

INTERVENTIONS:
Procedure: Breast Reconstruction, Direct to Implant (DTI) with Strattice™
  Arms: Breast Reconstruction, Direct to Implant (DTI) with Strattice™
Procedure: Two Stage Breast Reconstruction
  Arms: Two Stage Breast Reconstruction

SUMMARY:
The purpose of this study was to compare the efficacy of immediate single-stage post-mastectomy breast reconstruction with Strattice Reconstructive Tissue Matrix (Strattice) as compared to immediate two-stage post-mastectomy breast reconstruction where the initially placed expander was exchanged for a breast implant only, without any type of reinforcement.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the efficacy of immediate single-stage post-mastectomy breast reconstruction with Strattice™ TM, otherwise referred to as DTI as compared to immediate two-stage post-mastectomy breast reconstruction where the initially placed expander will be exchanged for a breast implant only, without any type of a reinforcement. The objective will be achieved by prospectively assessing the number of planned and unplanned post-mastectomy surgical interventions within 12 months of the mastectomy.

Two-stage breast reconstruction will include the initial placement of a tissue expander in a total or partial submuscular position. In the case of partial muscle coverage, this will be without the support of any mesh or autologous flap to reinforce the lower pole. The expander will be inflated over approximately the next one to six months, and then replaced with an implant.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years or older
* A candidate for both arms of the study involving immediate breast reconstruction post-skin sparing mastectomy (unilateral or bilateral) DTI with the use of Strattice™ Reconstructive Tissue Matrix (TM), 2 stage with use of Tissue Expander through exchange to Implant without support of a mesh or autologous tissue)
* An American Society of Anesthesiologists (ASA) Physical Status Classification of 1 or 2
* Estimated life expectancy > 3 years
* Able and willing to return for all scheduled and required study visits
* Able to provide written informed consent for study participation

Exclusion Criteria:

* Clinically significant systemic disease, as determined by the Investigator, which could affect study participation or study results
* Received neo-adjuvant, inductive chemo-therapy (except Herceptin, or other targeted therapy) within 4 weeks prior to mastectomy
* Previous radiation therapy to either breast at any time
* Predicted permanent implant size that is greater than or equal to 500 grams (gms), per Investigator assessment
* Body mass index (BMI) <17 or > 30
* Co-morbid factors which predispose to postoperative infection, e.g. diabetes, collagen vascular disease, chronic steroid (except inhalers)/immunosuppressant use, immune deficiency, or co-existent infection
* Pregnant or lactating
* 3rd degree ptosis
* Prior breast surgery including breast reduction, augmentation, mastopexy, quadrectomy, and partial mastectomy with reduction of the skin envelope
* Prior use of a device (mesh or matrix) in the Breast
* Concomitant unrelated condition of breast/chest wall/skin that, as determined by the investigator, could adversely affect the surgical outcome (e.g. significant chest wall abnormalities including pectus excavatum or pectus carinatum)
* Planned autologous tissue flap in addition to prosthetic implant
* Use of permanent expander implants such as Becker expanders or the Natrelle™ Permanent expander 150
* Current alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or drug abuse or addiction
* Currently enrolled or plans to enroll in another clinical trial unless it is: a registry, a retrospective study, a neo-adjuvant chemotherapy trial (as long as the chemotherapy regimen has been stopped 4 weeks prior to mastectomy), or a hormone/anti-hormonal therapy trial
* Any of the conditions identified within the labelled contraindications, i.e. sensitivity to porcine derived products or polysorbate 20.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Single Stage Breast Reconstruction in Female Participants with Mastectomy
Enrollment: 131 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Jacobs, Study Chair — Allergan
Locations (18):
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Institut du Cancer de Montpellier Val d'Aurelle, Montpellier
  - L'Institut du Sein- Paris Breast Center, Paris
  - Hopital Tenon APHP, Paris
- Germany (8):
  - Universitätsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitäts-Frauenklinik Heidelberg, Heidelberg
  - Klinik der Universität München, Campus Innenstadt, Munich
  - Klinikum rechts der Isar, Munich
  - Asklepios Paulinen Klinik, Wiesbaden
- United Kingdom (5):
  - St Luke's hospital / Bradford Royal Infirmary (BRI), Bradford
  - Dorset County Hospital, Dorchester
  - Frimley Park Hospital, Frimley
  - Wythenshawe Hospital UHSM NHS Foundation Trust, Manchester
  - City Hospital, Nottingham

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 131 enrolled participants, 127 received the study device and were included in the Safety population.
Period: Overall Study
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
Started | 76 | 55
Safety Set | 76 | 51 (4 participants did not have first surgery date and were not included in Safety Set.)
Completed | 71 | 23
Not Completed | 5 | 32
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Protocol Deviation | 0 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Study Terminated by Sponsor | 1 | 17
Not completed — Other Miscellaneous Reasons | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who underwent a mastectomy followed by one of the two implant-based breast reconstruction methods and had their first surgery date recorded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction | Total
Number analyzed (Participants) | 76 | 51 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (10.58) | 49.5 (10.40) | 47.9 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 51 | 127
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 1 | 0 | 1
  Caucasian | 51 | 35 | 86
  Other | 2 | 0 | 2
  Missing | 22 | 16 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Non-Hispanic or non-Latino | 53 | 34 | 87
  Missing | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Planned and Unplanned Post-mastectomy Surgical Interventions Per Participant on the Reconstructed Breast, Within 12 Months of the Initial Study Surgery (ISS)
Description: ISS was defined as the DTI breast reconstruction with Strattice™ or the first surgery of the two-stage breast reconstruction. Data is presented for participants with unilateral (one breast) and bilateral (two breast) reconstruction. Postmastectomy surgical interventions on the reconstructed breast were reported for each participant and the total number of planned and unplanned post-mastectomy surgical interventions was averaged in each group.
Time Frame: Up to 12 months post ISS
Population: Post-ISS analysis set consisted of all participants who underwent a mastectomy and completed their first reconstruction surgery post-mastectomy and have a valid surgical assessment at least 337 days post ISS (12 month [365 days]-4 week [28 days] window). Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: interventions per participant
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
Number analyzed (Participants) | 69 | 40
interventions per participant
  Unilateral: number analyzed (Participants) | 48 | 29
  Unilateral | 1.6 (1.87) | 2.2 (1.91)
  Bilateral: number analyzed (Participants) | 21 | 11
  Bilateral | 1.2 (1.99) | 2.3 (1.10)

2. Secondary Outcome: Number of Participants Experiencing One or More Serious Breast Reconstruction-related Complications (BRRC)
Description: Serious BRRC were complications that required re-entry of the breast pocket with or without exchange or removal of the implant and any manipulation of the implant pocket including the infra-mammary fold (IMF). Serious BRRC were detected through review by a medical monitor. Surgical complications included: capsular contracture (Baker grade ≥ 3), infection (local or systemic), hematoma, seroma, inflammation, skin or flap necrosis, implant extrusion, malposition, malrotation, asymmetry, bottoming out.
Time Frame: Up to 12 months post ISS
Population: Post-ISS analysis set consisted of all participants who underwent a mastectomy followed by one of the two implant-based breast reconstruction methods and completed their first reconstruction surgery post-mastectomy and have a valid surgical assessment at least 337 days post ISS (12 month [365 days]-4 week [28 days] window).
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
Number analyzed (Participants) | 69 | 40
Participants | 15 | 8

3. Secondary Outcome: Number of Participants Experiencing One or More Serious BRRC Within 24 Months of Post-Permanent Reconstruction (ppR)
Description: Serious BRRC were complications that required re-entry of the breast pocket with or without exchange or removal of the implant and any manipulation of the implant pocket including the IMF. Serious BRRC were detected through review by a medical monitor. BRRC were defined as: a) infection, local or systemic, b) hematoma, c) seroma, d) inflammation, e) skin or flap necrosis, f) capsular contraction as defined by Baker grade > 3, g) implant extrusion (loss or explants), and h) malposition, malrotation, asymmetry, and bottoming out.
Time Frame: Up to 24 months ppR
Population: ppR Follow-up set consisted of all participants who underwent a mastectomy followed by one of the two implant-based breast reconstruction methods and completed the 24 months ppR visit. Participants whose 24-month visit was performed early due to termination of the study were also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
Number analyzed (Participants) | 72 | 40
Participants | 19 | 9

4. Secondary Outcome: Number of Participants With Clinically Significant Cases of Capsular Contracture as Defined by Baker Grade III or IV Within 24 Months of ppR
Description: The surgeon assessed the level of capsular contracture in the participant's breast using the Baker Breast Contracture Scale where: Grade I=breast is normally soft and looks natural, Grade II=breast is a little firm but looks normal, Grade III=breast is firm and looks abnormal and Grade IV= breast is hard, painful, and looks abnormal. Baker Grade III and IV were defined as clinically significant and are reported here. Data is presented for number of participants with capsular contracture per breast (right breast and left breast).
Time Frame: Up to 24 months ppR
Population: Safety set included all participants who underwent a mastectomy followed by one of the two implant-based breast reconstruction methods and had their first surgery date recorded. Number analyzed for each category includes those participants for whom the Baker grade was assessed.
Measure: Number; unit: participants
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
Number analyzed (Participants) | 76 | 51
participants
  Right breast (Grade III): number analyzed (Participants) | 43 | 20
  Right breast (Grade III) | 0 | 0
  Right breast (Grade IV): number analyzed (Participants) | 43 | 20
  Right breast (Grade IV) | 0 | 0
  Left Breast (Grade III): number analyzed (Participants) | 48 | 24
  Left Breast (Grade III) | 1 | 0
  Left Breast (Grade IV): number analyzed (Participants) | 48 | 24
  Left Breast (Grade IV) | 0 | 0

5. Secondary Outcome: Aesthetic Outcomes of Participants Using Blinded Assessment 2D Photographs by Independent Review Panel
Time Frame: Baseline up to Month 24
Population: The independent reviewer panel was not established and data were not collected due to early termination of the study, hence this endpoint could not be analyzed.
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Planned and Unplanned Post-mastectomy Surgical Interventions of the Reconstructed Breast Within 6 Months of ISS
Description: as for outcome 1
Time Frame: Baseline up to 6 months post ISS
Population: Safety set included all participants who underwent a mastectomy followed by one of the two implant-based breast reconstruction methods and had their first surgery date recorded. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: interventions per participant
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
Number analyzed (Participants) | 76 | 51
interventions per participant
  Unilateral: number analyzed (Participants) | 53 | 36
  Unilateral | 1.1 (1.43) | 1.4 (1.40)
  Bilateral: number analyzed (Participants) | 23 | 15
  Bilateral | 1.0 (1.76) | 0.9 (1.28)

7. Secondary Outcome: Number of Planned and Unplanned Post-mastectomy Surgical Interventions of the Reconstructed Breast
Description: Surgical interventions were all planned and unplanned post-mastectomy surgical interventions per participant on the reconstructed breast, within 24 months of the ISS, which is defined as the DTI breast reconstruction with Strattice™ TM or the first surgery of the two-stage breast reconstruction. Data is presented for participants with unilateral (one breast) and bilateral (two breast) reconstruction.
Time Frame: Within 24 months ppR
Population: ppR Follow-up set included all participants who underwent a mastectomy followed by one of the two implant-based breast reconstruction methods and completed 24 months ppR visit; whose 24-month visit was performed early due to termination of study were also included. Number analyzed is number of participants with data available at given time-point.
Measure: Mean (Standard Deviation); unit: interventions per participant
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
Number analyzed (Participants) | 72 | 40
interventions per participant
  Unilateral: number analyzed (Participants) | 50 | 28
  Unilateral | 2.1 (2.04) | 3.0 (2.60)
  Bilateral: number analyzed (Participants) | 22 | 12
  Bilateral | 1.6 (2.42) | 2.8 (1.29)

8. Other Pre Specified Outcome: Health-related Quality of Life
Time Frame: At 3, 6, and 12 months post-mastectomy and at 4 months ppR
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Healthcare Resource Use Including Length of Hospital Stay and Clinic Visits
Time Frame: At 6 and 12 months post-mastectomy and at 24 months ppR
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Time to Return to Work or Normal Daily Activities
Time Frame: 6 and 12 months post-mastectomy and 24 month ppR
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first day post-surgery up to 24 months for participants enrolled in the Breast Reconstruction, DTI arm and approximately 25-30 months for participants enrolled in the Two-stage Reconstruction arm.
Description: The number of participants at risk for Serious Adverse Events and Other Adverse Events is based on the Safety Set. 4 participants did not have first surgery date and were not included in Safety Set.
Arm/Group | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ | Two Stage Breast Reconstruction
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/55
Serious Adverse Events (participants affected / at risk) | 49/76 | 27/51
Other Adverse Events (participants affected / at risk) | 53/76 | 35/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ (N=76) | Two Stage Breast Reconstruction (N=51)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Anisomastia (Reproductive system and breast disorders) | 5 | 3
Menorrhagia (Reproductive system and breast disorders) | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Capsular contracture associated with breast implant (Reproductive system and breast disorders) | 2 | 2
Mastoptosis (Reproductive system and breast disorders) | 0 | 1
Red breast syndrome (Reproductive system and breast disorders) | 1 | 0
Biopsy lymph gland abnormal (Investigations) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pyrexia (General disorders) | 2 | 0
Impaired healing (General disorders) | 2 | 0
Fat tissue decreased (General disorders) | 5 | 4
Medical device discomfort (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Device extrusion (Product Issues) | 3 | 1
Device dislocation (Product Issues) | 1 | 3
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Salpingo-oophorectomy (Surgical and medical procedures) | 0 | 2
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 | 2
Breast operation (Surgical and medical procedures) | 2 | 1
Mammoplasty (Surgical and medical procedures) | 1 | 0
Breast reconstruction (Surgical and medical procedures) | 12 | 1
Medical device removal (Surgical and medical procedures) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Device deployment issue (Injury, poisoning and procedural complications) | 1 | 0
Skin scar contracture (Injury, poisoning and procedural complications) | 2 | 0
Skin flap necrosis (Injury, poisoning and procedural complications) | 3 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 5 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 2 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 7 | 2
Breast cellulitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Breast Reconstruction, Direct to Implant (DTI) With Strattice™ (N=76) | Two Stage Breast Reconstruction (N=51)
Erythema (Skin and subcutaneous tissue disorders) | 10 | 8
Breast pain (Reproductive system and breast disorders) | 4 | 6
Capsular contracture associated with breast implant (Reproductive system and breast disorders) | 4 | 3
Breast inflammation (Reproductive system and breast disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 3
Fatigue (General disorders) | 1 | 4
Impaired healing (General disorders) | 5 | 1
Asthenia (General disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 4 | 6
Drug hypersensitivity (Immune system disorders) | 4 | 2
Device dislocation (Product Issues) | 0 | 3
Hot flush (Vascular disorders) | 4 | 5
Neuropathy peripheral (Nervous system disorders) | 1 | 3
Seroma (Injury, poisoning and procedural complications) | 26 | 13
Post procedural haematoma (Injury, poisoning and procedural complications) | 5 | 13
Wound secretion (Injury, poisoning and procedural complications) | 5 | 1
Procedural pain (Injury, poisoning and procedural complications) | 6 | 12
Wound dehiscence (Injury, poisoning and procedural complications) | 4 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 5
Mastitis (Infections and infestations) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.